CLINICAL TRIAL: NCT00276783
Title: A Phase II Trial of Alimta (Pemetrexed) in Patients With Recurrent Malignant Gliomas, Primary Central Nervous System Lymphoma, and Brain Metastases
Brief Title: Pemetrexed Disodium in Treating Patients With Recurrent Malignant Gliomas, Primary CNS Lymphoma, or Brain Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 05C2; P30CA060553 (NIH); NU-05C2; STU00007255 (Other: Northwestern University IRB)
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Brain and Central Nervous System Tumors; Lymphoma; Metastatic Cancer
Keywords: primary central nervous system lymphoma; tumors metastatic to brain; recurrent adult brain tumor; adult giant cell glioblastoma; adult gliosarcoma; adult mixed glioma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult glioblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Lymphoma; Neoplasm Metastasis; Brain Neoplasms; Glioblastoma; Gliosarcoma; Glioma; Astrocytoma; Oligodendroglioma | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Pemetrexed 900 mg/m2 every 21 days until disease progression.
  Interventions: Drug: pemetrexed

INTERVENTIONS:
Drug: pemetrexed — Administered intravenously at a dose of 900 mg/m2 every 21 days until disease progression.
  Other Names: pemetrexed disodium; Alimta

SUMMARY:
RATIONALE: Pemetrexed disodium may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well pemetrexed disodium works in treating patients with recurrent malignant gliomas, primary CNS lymphoma, or brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 6-month progression-free survival rate in patients with recurrent malignant gliomas treated with pemetrexed disodium.
* Determine the time to progression in patients with recurrent malignant gliomas, primary CNS lymphoma (PCNSL), or brain metastases treated with pemetrexed disodium.

Secondary

* Determine the radiographic response in patients with recurrent malignant gliomas, PCNSL, or brain metastases treated with pemetrexed disodium.
* Determine the time to response in patients treated with this drug.
* Determine the duration of response in patients treated with this drug.
* Determine the overall survival of patients treated with this drug.
* Collect safety data on patients with intracranial tumors treated with this drug.

OUTLINE: Patients receive pemetrexed disodium IV over 10 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 47 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Malignant glioma, including the following subtypes: glioblastoma or gliosarcoma, anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic mixed glioma, or malignant glioma not otherwise specified, meeting the following criteria:

    * Not required to have measurable or evaluable disease
    * Must have failed prior radiation therapy > 4 weeks ago
    * Must have failed at least 1 prior chemotherapy regimen
    * Confirmation of tumor progression by MR spectroscopy, PET scan, or biopsy/resection if prior radiosurgery was performed
  * Primary CNS lymphoma, meeting the following criteria:

    * Measurable disease as defined by bidimensionally measurable lesions with clearly defined margins by CT scan or MRI
    * Must have failed at least one prior chemotherapy regimen
    * Must have failed at least one agent or regimen
  * Brain metastases from a solid tumor, meeting the following criteria:

    * Measurable disease as defined by bidimensionally measurable lesions with clearly defined margins by CT scan or MRI
    * Biopsy is not required if radiographic imaging is consistent with brain metastases
    * Must have failed prior whole-brain radiotherapy
    * Patients with leptomeningeal metastases with or without brain metastases are eligible for therapy (may be diagnosed by MRI or cytology)
    * Confirmation of tumor progression by MR spectroscopy, PET scan, or biopsy/resection if prior radiosurgery was performed
* Effusions or fluid collections must be drained prior to study entry

PATIENT CHARACTERISTICS:

* Karnofsky performance score ≥ 60
* WBC > 3,000/mm^3
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 10 mg/dL (transfusion allowed)
* SGOT/SGPT < 3.0 times upper limit of normal (ULN)
* Bilirubin < 1.5 times ULN
* Creatinine < 1.5 mg/dL
* Creatinine clearance > 45 mL/min
* Women of childbearing potential and sexually active males must commit to the use of effective contraception while on study and for 3 months after completing study treatment
* Women who are pregnant or breast-feeding are not eligible for study treatment
* Negative pregnancy test
* Able to take steroids, vitamin B12, or folate
* No significant medical illnesses or infection that, in the investigator's opinion, cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy
* Only one active tumor type allowed, except nonmelanoma skin cancer or carcinoma in situ of the cervix

  * A history of other malignancies are acceptable if in complete remission and off all therapy for that disease for a minimum of 3 years

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior whole-brain or other radiotherapy
* Recovered from any side effects (6 weeks for a nitrosourea; 4 weeks for temozolomide, procarbazine, etoposide or experimental agent; 3 weeks for isotretinoin or tamoxifen) (for patients with gliomas)
* No more than 2 prior chemotherapeutic agents or regimens (includes biologic agents) (for patients with gliomas)
* Recovered from prior biopsy or re-resection of the tumor (10-14 days for resection or 3-5 days for a biopsy) (for patients with gliomas)
* May not be on any other chemotherapy except for hormonal therapy or trastuzumab (Herceptin®) (for patients with brain metastases)
* No limitations on prior CNS-directed therapies (for patients with brain metastases)
* Able to discontinue nonsteroidal anti-inflammatory drugs (NSAIDs)
* Patients taking NSAIDs or aspirin are required to interrupt therapy for at least 2 days before the study treatment and 2 days after the infusion

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-11; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival at 6 months and time to disease progression | After every 2 cycles of therapy (1 cycle = 3 weeks) until disease progression

SECONDARY OUTCOMES:
Radiographic response | After 6 months of treatment
Collect safety data | After every cycle of therapy (cycle = 3 weeks) until disease progression or death.
Overall survival | After every cycle of treatment (1 cycle = 3 weeks) until death
Compare blood and tissue methylation patterns and correlate with response. | Blood and tissue from baseline, then additional blood every 6 weeks while on treatment
  This was optional for patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J. Raizer, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (2):
- United States (2):
  - Hematology-Oncology Associates of Illinois, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois